CLINICAL TRIAL: NCT00634673
Title: FABP2 Ala54Thr Genotype Influences the Postprandial Serum Fatty Acids Profile in Type 2 Diabetic Patients
Brief Title: Postprandial Fatty Acids and FABP2 in Type 2 Diabetes Mellitus (DM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: MIrela Jobim de Azevedo, Hospital de Clínicas de Porto Alegre
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: HCPA05060
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-02

CONDITIONS: Dyslipidemia; Type 2 Diabetes Mellitus
Keywords: Serum Fatty Acids; FABP2 Gene; Polymorphism Ala54Thr
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TT (Other): patients homozygous for Thr54 (TT)
  Interventions: Other: sandwich
- AA (Other): patients homozygous for Ala54 (AA)
  Interventions: Other: sandwich

INTERVENTIONS:
Other: sandwich — standard meal:sandwich (7.23 kcal/kg-total energy; 43.35% fat, 21.95% protein, and 34.70% carbohydrate)
  Other Names: fat meal

SUMMARY:
This study will be conducted in type 2 diabetic patient's to evaluate the if there is a different response of serum lipids after a standard meal (rich in saturated fatty acids) in patients who have the presence of a genetic alteration. This alteration that will be evaluated is a polymorphism, change of an amino acid in the gene of FABP2. This gene that can influence the absorption of lipids in the intestine and subjects who have the altered genotype (presence of T allele) can have an abnormal lipid profile as compared to subjects without this genotype.

DETAILED DESCRIPTION:
Background: The presence of Ala54Thr polymorphism of intestinal fatty acid-binding protein 2 gene (FABP2) might influence the intestinal absorption of dietary fatty acids (FAs) and has been associated with diabetic nephropathy.

Objective: We studied the postprandial serum FAs in type 2 diabetic patients homozygous for Thr54 (TT; n = 11) or for Ala54 (AA; n = 15) after a standard meal.Design: Patients received a sandwich (7.23 kcal/kg-total energy; 43.35% fat, 21.95% protein, and 34.70% carbohydrate) in the morning after 12-h fasting and FAs in chylomicrons (gas chromatograph), plasma glucose, and serum triacylglycerols were measured at 0, 2, 4, 6 and 8 h. Results: TT and AA patients did not differ regarding age (61.6±6.7 vs. 62.0±7.7years), diabetes duration (12.7±6.9 vs. 13.1±5.6years), male proportion (72.7 vs. 86.7%), blood pressure, type of diabetes treatment and previous macronutrients intake as well as serum A1C test (6.5±0.6 vs. 6.7±0.4%), LDL (3.0±1.0 vs. 3.2±0.6mmo/L), HDL (1.3±0.2 vs. 1.3±0.4mmol/L), triacylglycerols [1.6(1.0-3.4) vs. 1.6(0.6-3.7)mmol/L], saturated, monounsaturated, and polyunsaturated FAs, and trans-unsaturated FAs. The increase in serum glucose and triacylglycerols after the meal (ANOVA,P<0.001) was not different in both groups. The maximum increase of FAs occurred at 6-h postprandial, but only in TT patients: saturated FAs increased from 464.4(56.9-1602.5) to 1249.5(214.5-7149.8)mg/dL (P=0.041), monounsaturated FAs from 387.9(30.2-1523.8) to 925.1(344.6-5554.0)mgd/L (P=0.026), polyunsaturated FAs from 258.9(0-1048.5) to 713.1(143.7-7987.6)mg/dL (P=0.021), trans-unsaturated FAs from 18.5(1.9-70.6) to 66.5(5.0-451.7)mg/dL (P=0.023). Conclusion: The presence of the T allele of Ala54Thr polymorphism of FABP2 gene in type 2 diabetic patients increases absorption of dietary FAs, including the trans-unsaturated FAs, and this might turns these patients more susceptible to the effect of diet composition.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* homozygote to FABP2 polymorphism:TT or AA

Exclusion Criteria:

* age >75 years
* glomerular filtration rate <30ml min-1
* with unstable angina or possible infarct or stroke in the last year

Ages: 40 Weeks to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
postprandial serum fatty acids | 0, 2, 4,6, and 8 hours after meal

SECONDARY OUTCOMES:
serum endothelin serum fibrinogen | 0 and 8 hours after meal

CONTACTS AND LOCATIONS:
Overall Officials: Mirela J Azevedo, MD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Almeida JC, Gross JL, Canani LH, Zelmanovitz T, Perassolo MS, Azevedo MJ. The Ala54Thr polymorphism of the FABP2 gene influences the postprandial fatty acids in patients with type 2 diabetes. J Clin Endocrinol Metab. 2010 Aug;95(8):3909-17. doi: 10.1210/jc.2009-2674. Epub 2010 May 19. PMID 20484485